CLINICAL TRIAL: NCT01523938
Title: Influence of Perioperative Hypnotherapy on Postoperative Improvement in Cognitive Performance. A Randomized-controlled Open Clinical Monocentric Interventional Study.
Brief Title: Influence of Perioperative Hypnotherapy on Postoperative Improvement in Cognitive Performance
Acronym: HYPNOC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Prof., MD Director of the Department of Anaesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYPNOC
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Hypnotherapy
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnotherapy (Experimental)
  Interventions: Behavioral: Hypnotherapy
- No Hypnotherapy (No Intervention)

INTERVENTIONS:
Behavioral: Hypnotherapy — Pre- (one session) and postoperative (two sessions) Hypnotherapy
  Arms: Hypnotherapy

SUMMARY:
The study examines prospects of hypnotherapy in reducing agitation in patients after cardiac or spinal column surgery. A particular aim is to point out the effects on postoperative cognitive outcome. Additional blood and urine tests are conducted (concerning cardiac stratum).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients scheduled for open heart surgery or spinal column surgery
* Offered patient information and written informed consent
* Mini Mental State > 23
* American Society of Anesthesiologists physical status classification system (ASA) 1-3

Exclusion Criteria:

* No informed consent
* Patients aged <18 years
* Patients living outside Berlin/Potsdam and surrounding area
* Less than 5 points in Stanford Scale of Hypnotic Susceptibility: Form C; German version (SHSS:C -Weitzenhoffer & Hilgard, 1962; Bongartz, 1999 a)in the screening/recruiting phase
* Lacking consent capability or accommodation in an institution due to an official or judicial order
* Emergency patients or ambulant patients
* Pregnancy and lactation
* Coworkers at Charité
* Lacking willingness to save and hand out data within the study
* Insufficient knowledge of the German language
* Participation in another trial according to the German Drug Law the week before inclusion (in the study) and the parallel participation in another trial according to the German Drug Law within the first 3 months after surgery
* Acute, severe psychic disease (acute psychotic disorder, severe drug dependency, withdrawal symptoms)
* Conditions which make a sufficient information and consequent consent impossible
* The patient is under juridical supervision
* acute risk of suicide
* dementia
* patients who suffer from insulin dependent Diabetes mellitus and who have been diagnosed with Diabetes mellitus within the last year
* patients who have suffered allergic shock in the past
* hardness of hearing, deafness, blindness
* cardiac function: ejection fraction (EF) < 30%
* Patients undergoing psychotherapeutic treatment
* Patients taking awareness-modulating drugs (antipsychotic drugs)
* Boozed/primed patients or patients under drug influence
* Patients having had an epileptic seizure within the last four weeks
* Patients suffering from productive cough
* Patients having a chronic low blood pressure (systolic <90mmHg)
* Allergies to any ingredient of the electrode fixing material (only for participants of sleep stage assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction at the time of discharge | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).

SECONDARY OUTCOMES:
Incidence of postoperative cognitive dysfunction three months after surgery | three months after surgery
Postoperative delirium | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction in pre- and postoperative agitation and anxiety | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction of pain | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction of stress | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction of holding time | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction of hospital stay | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Reduction of Intensive Care Unit stay | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Readmission rate | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Emotional status | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery).
Functional status | on day 7 - 30 after surgery
  Planned measures on the seventh postoperative day or on day of hospital discharge (≤ 30 days after surgery)
Subjective evaluation of sleep quality | Before surgery
  Insomnia Severity Index (ISI)
Perioperative assessment of sleep stage | the night after surgery;the night before discharge; 3 months after surgery

OTHER OUTCOMES:
Additional blood and urine tests (concerning cardiac stratum) | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  * oxidized Parathyroid hormone and real intact, biologically active Parathyroid hormone
  * Urine: Creatinin, ionized Calcium, Phosphate
  * Calprotectin
  * S100A12
  * Arterial blood: Calcium ionized, Phosphate and potential of hydrogen (pH)
  * 3-hydroxy-3-methyl-glutaryl-CoA reductase
  * Mevalonate
  * Procalcitonin

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Department of Anaesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum (CVK) and Campus Charite Mitte (CCM), Charite - Universitätsmedizin Berlin
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum (CVK) and Campus Charite Mitte (CCM), Charite - Universitätsmedizin, Berlin, State of Berlin, Germany